CLINICAL TRIAL: NCT01141465
Title: A Retrospective Evaluation of the Effectiveness of Fixed-dose Combination Inhaled Corticosteroid /. Long-acting Beta Agonist (ICS/LABA) Therapy in the Management of Asthma in a Representative UK Primary Care Population
Brief Title: Real-world Effectiveness of Combination Therapy in Asthma
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Mundipharma Research Limited (Industry)
Responsible Party: Professor David Price, Research in Real Life Limited
Other Study IDs: BS30
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Asthma
Keywords: Primary care; Asthma management; Combined therapy; Real-world; Effectiveness; Control; Exacerbations
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Budesonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- IPDA FP/SAL DPI: Patients who were on inhaled corticosteroid therapy during the baseline year (any ICS therapy) who, at an index prescription date, initiated combination therapy as FP/SAL DPI at ≥twice the equivalent BDP-equivalent dose
  Interventions: Drug: Fluticasone / salmeterol dry powder inhaler
- IPDA FP/SAL MDI: Patients who were on inhaled corticosteroid therapy during the baseline year (any ICS therapy) who, at an index prescription date, initiated combination therapy as FP/SAL MDI at ≥twice the equivalent BDP-equivalent dose
  Interventions: Drug: Fluticasone / salmeterol metred dose inhaler
- IPDI FP/SAL DPI: Patients who were on inhaled corticosteroid therapy during the baseline year (any ICS therapy) who, at an index prescription date, initiated combination therapy as FP/SAL DPI at equivalent BDP-equivalent dose
  Interventions: Drug: Fluticasone / salmeterol dry powder inhaler
- IPDI BUD/FOR DPI: Patients who were on inhaled corticosteroid therapy during the baseline year (any ICS therapy) who, at an index prescription date, initiated combination therapy as BUD/FOR DPI at equivalent BDP-equivalent dose
  Interventions: Drug: Budesonide / formoterol dry powder inhaler
- IPDI FP/SAL MDI: Patients who were on inhaled corticosteroid therapy during the baseline year (any ICS therapy) who, at an index prescription date, initiated combination therapy as FP/SAL MDI at equivalent BDP-equivalent dose
  Interventions: Drug: Fluticasone / formoterol metered dose inhaler
- IPDA BUD/FOR DPI: Patients who were on inhaled corticosteroid therapy during the baseline year (any ICS therapy) who, at an index prescription date, initiated combination therapy as BUD/FOR DPI at ≥twice the equivalent BDP-equivalent dose
  Interventions: Drug: BUD/FOR dry powder inhaler

INTERVENTIONS:
Drug: Fluticasone / formoterol metered dose inhaler — Prescribed at the same BDP-equivalent dose as baseline ICS
  Other Names: Seretide MDI
  Groups: IPDI FP/SAL MDI
Drug: Fluticasone / salmeterol dry powder inhaler — Prescribed at the same BDP-equivalent dose as baseline ICS
  Other Names: Seretide DPI
  Groups: IPDI FP/SAL DPI
Drug: Budesonide / formoterol dry powder inhaler — Prescribed at the same BDP-equivalent dose as baseline ICS
  Other Names: Symbicort DPI
  Groups: IPDI BUD/FOR DPI
Drug: Fluticasone / salmeterol dry powder inhaler — Prescribed at ≥twice BDP-equivalent dose as baseline ICS
  Other Names: Seretide DPI
  Groups: IPDA FP/SAL DPI
Drug: Fluticasone / salmeterol metred dose inhaler — Prescribed at ≥twice BDP-equivalent dose as baseline ICS
  Other Names: Seretide MDI
  Groups: IPDA FP/SAL MDI
Drug: BUD/FOR dry powder inhaler — Prescribed at ≥twice BDP-equivalent dose as baseline ICS
  Other Names: Symbicort DPI
  Groups: IPDA BUD/FOR DPI

SUMMARY:
This study will evaluate and compare the effectiveness of asthma management in patients with evidence of persistent asthma following a switch in asthma therapy to combination inhaled glucocorticosteroid (ICS) / long-acting bronchodilator (LABA) therapy as either: fixed-combination fluticasone propionate / salmeterol (FP/SAL; Seretide®) via pressurised metered-dose inhaler (pMDI) or dry-powder inhaler (DPI) plus as-needed (prn) reliever therapy (salbutamol as DPI, BAI or pMDI), or fixed-combination budesonide / formoterol (BUD/FOR; Symbicort®) via DPI plus prn reliever therapy (salbutamol as DPI, BAI or pMDI or bricanyl as DPI). The final analysis plan will define exact comparators and age groups to be studied after reviewing baseline data.

DETAILED DESCRIPTION:
Current asthma guidelines in the UK are underpinned by evidence derived from randomised controlled trials (RCTs). Although RCT data are considered the gold standard, patients recruited to asthma RCTs are estimated to represent less than 10% of the UK's asthma population. The poor representation of the asthma population is due to a number of factors, such as tightly-controlled inclusion criteria for RCTs. There is, therefore, a need for more representative RCTs and real-life observational studies to inform existing guidelines and help optimise asthma outcomes.

The fixed combination asthma inhalers FP/SAL (as pMDI and DPI) and BUD/FOR (as DPI) are indicated for use in asthma when adequate asthma control is not achieved with low / medium dose ICS therapy and prn reliever therapy (a short-acting beta-agonist [SABA]). Fixed combination inhalers are also indicated in patients already adequately controlled on separate ICS/LABA therapy. However, emerging trends in asthma prescribing indicate increasing use of add-on therapies (particularly in the form of combination inhalers) in the early stages of asthma therapy, even as first-line therapy.

The British Thoracic Society (BTS) Scottish Intercollegiate Guidelines Network (SIGN) guidelines on the management of asthma advise that there is no difference in efficacy between ICS/LABA therapy given as separate or combined inhalers. However, they do note that, once a patients is on stable therapy, combination inhalers have the advantage of guaranteeing that patients do not take their LABA without their ICS.

In practice, there is significant pressure (supported by asthma guidelines) to use the least expensive, effective inhaled therapies available. While the effect of increased use of combination therapies in terms of patient benefits remains uncertain, the impact on treatment costs for the United Kingdom's (UK's) National Health Service (NHS) is unequivocal and, to date, there are limited data available as to the absolute and relative effectiveness of the ICS/LABA combination therapies currently licensed.

There are a number of inhaler delivery devices available for use in asthma management. Whatever therapy is prescribed, optimal treatment response requires effective drug delivery within the airways; selecting the most appropriate delivery device for an asthma patient, therefore, plays an important role in optimising their asthma control. According to the recent BTS/SIGN guidelines, there is currently no evidence of a clinical difference in the effectiveness of therapy delivery via pMDI ± spacer compared with DPI in either adults or children, and more recent DPIs are rated as effective as older DPIs. Effective use of DPIs and pMDI requires entirely different inhalation techniques and there is some debate as to whether patients prescribed different device types for their reliever and preventer medication (requiring different techniques for each) may have poorer disease control than those prescribed the same device type for both preventer and reliever. Combining aerosols (e.g. pMDI preventer plus BAI reliever) is not considered to cause a problem in this respect.

The aim of this study is to compare the absolute and relative effectiveness of currently licensed ICS/LABA combinations - FP/SAL and BUD/FOR (and their available delivery devices) - in children and adults with asthma whose therapy was changed or increased. Consideration will also be given to the effect of reliever therapy inhaler and the effect of consistency of device used (i.e. same or different devices for preventer and inhaler therapies) on asthma control outcomes. Also to be evaluated are the associated impact of inhaler technique review, recorded inhaler handling problems and use of a spacer in conjunction with a pMDI in terms of achieving asthma control outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 4-80 years: Paediatric cohort (aged 4-11 years); Adult cohort (aged 12-69 years); Elderly cohort (aged 70-80 years.
* Evidence of asthma: i.e. a diagnostic code of asthma or ≥2 prescriptions for asthma at different points in time during the prior year, including one ICS prescription.
* Be on current asthma therapy: i.e. ≥1 asthma prescriptions in the prior year, and at least 1 other asthma prescription during the same period.
* Have at least one year of up-to-standard (UTS) baseline data (prior to the IPD) and at least one year of UTS outcome data (following the IPD).

Exclusion Criteria:

* Diagnostic read code for chronic respiratory disease (including COPD) at any time
* On maintenance oral steroid therapy at baseline
* Any patients receiving a combination inhaler in addition to their separate ICS inhaler in the baseline year.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care asthma patients receiving ICS therapy (any of BDP, extrafine HFA-BDP, BUD or FP as pMDI, BAI or DPI) plus as needed SABA reliever therapy who underwent a change in asthma therapy to combination ICS/LABA therapy as FP/SAL (MDI or DPI) or BUD/FOR (DPI) at the same or at least twice the BDP-equivalent dose of ICS prescribed during baseline.
Sampling Method: Non-Probability Sample
Enrollment: 815377 (Actual)
Dates: Start 2001-01; Primary Completion 2007-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Composite proxy for asthma control | One-year outcome period
  * No recorded hospital attendance for asthma, including admission, Accident & Emergency (A&E) attendance, out-of-hours attendance, or Out-Patient Department (OPD) attendance, AND
  * No prescriptions for oral steroids, AND
  * No GP consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics.
Exacerbations (total and rate ratio) | One-year outcome period
  * Unscheduled hospital admissions / A&E attendance for asthma, AND/OR
  * Use of oral steroids.
GOAL Total Control (proxy measure to replicate total control as measured in the GOAL RCT in a real world patient population | 6 months (sensitivity analysis at 8 weeks)
  * No day-time symptoms;
  * No night-time symptoms;
  * No exacerbations;
  * No treatment-related adverse events
  * PEF ≥80% predicted = "normal"
  * No SABA use
GOAL exacerbations | One year
  Absence of:
  * Documented episodes of hospitalisations AND/OR
  * Exacerbation treatment - oral steroids or antibiotics for asthma over one year

SECONDARY OUTCOMES:
Compliance with ICS/LABA combination therapy | One year outcome period
  Percentage compliance calculated based on prescription refills
Compliance with ICS as part of ICS/LABA combination therapy | One-year outcome period
  Percentage compliance calculated based on prescription refill
Treatment success | One-year outcome period
  Success of the therapeutic regimen, defined as the absence of:
  * Exacerbation, and
  * Increased dose of ICS, and
  * Change in ICS/LABA, and
  * Change in delivery device, and
  * Use of additional therapy as defined by: oral steroids, theophylline, leukotreine receptor antagonists (LTRAs).
SABA dosage | One-year outcome period
  Categorised average SABA dosage during outcome year: 0mcg, >0-100mcg, >100-200mcg, >200-400mcg, >400-800mcg, >800mcg.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof. MD, Principal Investigator — Company Director; Alison Chisholm, MSc, Study Director — Research Project Director
Locations (1):
- General Practice Research Database, London, United Kingdom

REFERENCES:
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Travers J, Marsh S, Caldwell B, Williams M, Aldington S, Weatherall M, Shirtcliffe P, Beasley R. External validity of randomized controlled trials in COPD. Respir Med. 2007 Jun;101(6):1313-20. doi: 10.1016/j.rmed.2006.10.011. Epub 2006 Nov 17. PMID 17113277
- [Background] Appleton SL, Adams RJ, Wilson DH, Taylor AW, Ruffin RE; North West Adelaide Cohort Health Study Team. Spirometric criteria for asthma: adding further evidence to the debate. J Allergy Clin Immunol. 2005 Nov;116(5):976-82. doi: 10.1016/j.jaci.2005.08.034. PMID 16275363
- [Background] Bateman ED, Boushey HA, Bousquet J, Busse WW, Clark TJ, Pauwels RA, Pedersen SE; GOAL Investigators Group. Can guideline-defined asthma control be achieved? The Gaining Optimal Asthma ControL study. Am J Respir Crit Care Med. 2004 Oct 15;170(8):836-44. doi: 10.1164/rccm.200401-033OC. Epub 2004 Jul 15. PMID 15256389
- [Background] British Thoracic Society (BTS) Scottish Intercollegiate Guidelines Network (SIGN) 101. British Guideline on the Management of Asthma: a national clinical guideline. 2008. Available online at: www.sign.ac.uk/guidelines/fulltext/101/index.html
- See also: Optimum Patient Care is the Research in Real Life's sister company (a social enterprise organisation) — http://www.optimumpatientcare.org